CLINICAL TRIAL: NCT02158598
Title: Comparison of Changes in Serum 25(OH)D Concentrations Following Vitamin D Supplementation With Chewable Tablets Versus Pills
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Khlôros Technology (Unknown); Anne-Sophie Morisset (Unknown)
Responsible Party: Principal Investigator, Claudia Gagnon, MD, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B14-03-1896
Record Dates: First submitted 2014-06-02; First posted 2014-06-09 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D; Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- wash-out (No Intervention): 2 months
- Vitamin D chewable tablet supplementation (Experimental): A chewable vitamin D tablet containing 1000 IU to be taken once a day for 2 months.
  Interventions: Drug: Vitamin D chewable tablet supplementation
- Vitamin D pill supplementation (Experimental): A vitamin D pill containing 1000 IU to be taken once a day for 2 months.
  Interventions: Drug: Vitamin D pill supplementation

INTERVENTIONS:
Drug: Vitamin D chewable tablet supplementation
  Arms: Vitamin D chewable tablet supplementation
Drug: Vitamin D pill supplementation
  Arms: Vitamin D pill supplementation

SUMMARY:
This is a 6-month cross-over trial of vitamin D supplementation in 38 healthy men and women aged 18 years and older. The primary aim is to compare the change in serum 25(OH)D concentration following vitamin D supplementation with chewable tablets versus pills. Secondary aims are to evaluate satisfaction and adherence to the vitamin D chewable tablet supplement. Questionnaires on physical activity, sunlight exposure and dairy product consumption will be administered to adjust for confounding factors. A questionnaire will be administered to assess satisfaction and pill count to evaluate adherence to treatment. This research intends to test the hypothesis that the vitamin D chewable tablet supplement is as effective as a traditional vitamin D pill supplement to increase serum 25(OH)D concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men and women;
* Aged 18 years and older;
* Having a serum 25(OH)D concentration of 75 nmol/L or less.

Exclusion Criteria:

* Regular consumption of a supplement containing > 400 IU/d of vitamin D over the last 2 months;
* Intestinal malabsorption;
* Cirrhosis;
* Renal insufficiency (creatinine clearance <60 ml/min);
* Hypercalcemia;
* Pregnancy;
* Breastfeeding;
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-06; Primary Completion 2017-12 (Actual); Study Completion 2018-05-09 (Actual)

PRIMARY OUTCOMES:
Change in Serum 25(OH)D concentration | 0 and 2 months, 4 and 6 months

SECONDARY OUTCOMES:
Satisfaction with the vitamin D chewable tablets and pills. | 0 and 2 months, 4 and 6 months
  Satisfaction will be assessed using a questionnaire administered by the research team.
Adherence to the vitamin D chewable tablets and pills. | 0 and 2 months, 4 and 6 months
  This issue will be assessed by pill count.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Gagnon, MD, Principal Investigator — CHU de Québec Research Centre and Laval University
Locations (1):
- CHU de Québec Research Centre, Laval University, Québec, Quebec, Canada